CLINICAL TRIAL: NCT04365231
Title: Efficacy Evaluation of Hydroxychloroquine Azithromycin in the Treatment of COVID-19 in Pregnant Women: an Open-label Randomized Clinical Trial
Brief Title: Hydroxychloroquine Azithromycin COVID-19 Pregnancy Trial
Acronym: HASCOPT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no authorization obtained
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HASCOPT2020
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: COVID19
Keywords: SARS-Cov-2 virus; coronavirus disease; COVID-19; epidemic; pregnancy; RT-PCR; hydroxychloroquine; azithromycin; respiratory distress
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine and azithromycin treatment (Experimental): hydroxychloroquine 10-day course of hydroxychloroquine 200 mg tablet three times a day. To be taken orally.
  - azithromycin 5-day course of azithromycin 250 mg tablet twice a day on the first day of treatment, then once a day the 4 following days.
  Interventions: Drug: Hydroxychloroquine and azithromycin treatment; Other: conventional management of patients
- conventional management of patients (Active Comparator): Regular management of patients
  Interventions: Other: conventional management of patients

INTERVENTIONS:
Drug: Hydroxychloroquine and azithromycin treatment — hydroxychloroquine 10-day course of hydroxychloroquine 200 mg tablet three times a day. To be taken orally.
  - azithromycin 5-day course of azithromycin 250 mg tablet twice a day on the first day of treatment, then once a day the 4 following days.
  Arms: Hydroxychloroquine and azithromycin treatment
Other: conventional management of patients — conventional management of patients

SUMMARY:
Up to date, and since December 31st 2019, 2 520 522 cases of COVID-19 including 176 786 deaths, have been reported worldwide. Global efforts are made to save lives and decrease morbidity by evaluating therapeutic strategies. Pregnant women with COVID-19 are at high-risk of severe complications and mortality from COVID-19 infection, due to physiologic and immune changes occurring during pregnancy. These risks include development of maternal hypoxemic respiratory failure due to severe pneumonia, hospitalization in intensive care, death; but also, fetal morbidity-mortality with chronic and/or acute fetal distress, intrauterine growth retardation, intrauterine death and neonatal morbidity, mainly due to induced preterm birth and maternal-fetal transmission. Knowledge of these epidemiologic facts on SARS-Cov-2 infection in pregnant women is currently limited to small case-series. No drug has demonstrated solid evidence in treating SARS-Cov-2 virus. Nevertheless, in vitro studies and tests in COVID-19 positive patients treated with hydroxychloroquine and azithromycin merit further evaluation. Pregnant women are systematically excluded from drug trials, and treatment options for this high-risk population remain untested. The aim of this study is to screen pregnant women presenting minor symptoms, for COVID-19 and to evaluate efficacy of hydroxychloroquine-azithromycin treatment in preventing aggravation of symptoms with development of hypoxemic respiratory failure and complications of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* 18 and over
* monofetal pregnancy between 22+0 and 41+0 weeks of gestation
* presenting a positive COVID-19 RT-PCR test result after nasopharyngeal swab for one or more minor symptoms: cough, body temperature >37,3 °C, shortness of breath, diarrhea, asthenia, anosmia, taste loss, myalgia
* presenting no contraindication to hydroxychloroquine and azithromycin
* informed consent signature
* affiliated to social security scheme

Exclusion Criteria:

* allergic to hydroxychloroquine or chloroquine, or azithromycin
* contraindication to hydroxychloroquine: retinopathy, G6PD deficiency, long QT syndrome, any other heart rhythm abnormality on pre-recruitment electrocardiogram, hypokalemia, porphyria, psoriasis.
* contraindication to azithromycin: long QT syndrome, liver failure, myasthenia
* receiving simultaneous treatments contraindicated in case of hydroxychloroquine uptake: Citalopram (Seropram), escitalopram (Seroplex), hydroxyzin (Atarax), domperidone (Motilium), piperaquine (Eurartesim), disopyramide (Isorythm, Rythmodan), hydroquinidine chlorydrate (Serecor), amiodarone (Cordarone), dronedaron (Multaq), tricyclic antidepressant, anti-infectious drugs (macrolids, fluoroquinolones, trimethoprime-sulfamethoxazole (Bactrim).
* receiving simultaneous treatments contraindicated in case of azithromycin uptake: Cisapride, Colchicine, Dihydroergotamine, bromocriptine, cabergoline, lisurid, pergolide, atorvastatin, ciclosporin, digoxin, simvastatin, anti-vitamine K, macrolids, ketolide
* hypoxemic respiratory failure due to severe pneumonia (needing supplemental oxygen)
* maternal disorders: Type I or II diabetes, congenital cardiopathy, liver or kidney disease, liver failure, renal failure
* obstetrical disorders: insulin-dependent gestational diabetes, preterm delivery threat, preterm rupture of membranes, bleeding, pre-eclampsia, gestational hypertension, gestational cholestasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a negative RT-PCR test result to COVID-19 | 7 days
  Percentage of patients with a negative RT-PCR test result to COVID-19 nasopharyngeal swab at the 7th day of treatment by hydroxychloroquine and azithromycin.

SECONDARY OUTCOMES:
Maternal outcomes: Percentage of severe forms of the disease | 25 weeks
  percentage of severe forms of the disease
Newborn outcomes: Rate of newborns hospitalized in intensive care or transferred to resuscitation unit | 25 weeks
  rate of newborns hospitalized in intensive care or transferred to resuscitation unit

IPD SHARING:
Plan to Share IPD: No